CLINICAL TRIAL: NCT00226239
Title: A Phase II Trial of Docetaxel, Cetuximab (C225), and Cisplatin Followed by Radiation, Cetuximab, and Cisplatin in Locally Advanced Head and Neck Cancer
Brief Title: Docetaxel, Cetuximab and Cisplatin Followed by Radiation, Cetuximab and Cisplatin in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-003
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: head; neck
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel; Cisplatin; Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Head and neck cancer patients (Experimental): Induction chemotherapy consists of 3 cycles of cisplatin 75 mg/m^2, on day 1, docetaxel 75 mg/m^2, on day 1, and cetuximab weekly days 1,8,15, repeated every 21 days (cetuximab dose is 400 mg/m^2 on day 1 and 250 mg/m^2 on subsequent weekly treatments). After 3 cycles of induction, patients receive standard radiation 70 Gy/200 cGy/daily, 5 days/week with concurrent weekly cisplatin 30 mg/m^2 and cetuximab 250 mg/m^2. After completing radiation therapy, patients receive cetuximab weekly as maintenance therapy for 6 months (see section 5 for detailed treatment plan and dose modifications)
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Cetuximab; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m^2 IV over 1 hour, day 1
Drug: Cisplatin — Cisplatin 75 mg/m^2 IV over 1-2 hours, day 1, 1 hour following completion of cetuximab infusion.
Drug: Cetuximab — Cetuximab dose will be 250 mg/m^2 IV over 60 minutes weekly on ALL subsequent administrations (days 8 and 15 of cycle 1 and days 1,8,15 of cycles 2 and 3).
  Other Names: (Erbitux or C225)
Procedure: Radiation Therapy — Photon energies of 1.25 to 6 MV and/or appropriate electron energies for boosting the nodes are allowed. Photon energies>6 MV may be utilized when appropriate to boost target localized centrally.

SUMMARY:
The purpose of this study is to determine if the addition of a unique targeted agent called Cetuximab (also known as "C225" and "Erbitux") can increase the effectiveness of standard treatment with chemotherapy and radiation.

DETAILED DESCRIPTION:
This research study involves the use of a combination of two chemotherapies, cisplatin and docetaxel, which have been known to shrink head and neck cancers and are a commonly used treatment for this type of cancer. This combination will then be followed by radiation and more chemotherapy.

The purpose of this study is to see whether this combination of chemotherapy and radiation, with the addition of Cetuximab, can improve control of disease and collect information on what side effects this combination therapy may have. In addition, biologic factors (markers) will be studied that may help to predict and treat head and neck cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Stage III-IVB head and neck cancer, all sites, including unknown primary tumors (bulky stage II (T2N0) lesions of the base of tongue or hypopharynx and patients with stage II nasopharyngeal cancer are also eligible) Prior to study entry the resectability and alternative treatment options will be determined by a team composed of an Ear, Nose, and Throat Surgeon, a Radiation Oncologist and a Medical Oncologist. Stage determination, optimal local treatment, and its timing according to this protocol will be determined at this evaluation. Unequivocal demonstration of distant metastasis (M1) confers ineligibility
2. Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas, or WHO types I-III of the nasopharynx
3. Unidimensionally-measurable disease is required (RECIST)
4. No prior chemotherapy, biologic/molecular targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer
5. Prior surgical therapy will consist only of incisional or excisional biopsy and organ sparing procedures such as debulking of airway compromising tumors or neck dissection in a patient with an existing primary tumor (Any non-biopsy procedure must have taken place > 4 weeks but < 3 months of initiating protocol treatment)
6. ECOG PS 0 or 1; 7. Organ & marrow function per protocol criteria and 8. Age of >=18 years

Exclusion Criteria:

1. History of severe allergic reactions attributed to docetaxel or compounds of similar chemical or biologic composition to docetaxel, or other drugs formulated with polysorbate 80
2. Uncontrolled intercurrent illness or significant history of uncontrolled cardiac disease
3. Receiving any other investigational agents
4. No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, or malignancy that has been treated with a curative intent with a 5-year disease-free survival
5. Significant baseline sensory or motor neurologic deficits (> grade I neuropathy); 6. HIV-positive patients and 7. Prior severe infusion reaction to a monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bauman, MD, Principal Investigator — Univ of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Groups:
- Head and Neck Cancer Patients: Patients with locally advanced HNC, including squamous and undifferentiated histologies, treated with docetaxel 75 mg/m^2 day 1, cisplatin 75 mg/m^2 day 1, and cetuximab 250 mg/m^2 days 1, 8, and 15 (after an initial loading dose of 400 mg/m^2), termed TPE, repeated every 21 days for three cycles, followed by radiotherapy with concurrent cisplatin 30 mg/m^2 and cetuximab weekly (XPE), and maintenance cetuximab for 6 months.
Period: TPE, Induction Therapy
Arm/Group | Head and Neck Cancer Patients
Started | 39
Completed | 37
Not Completed | 2
Period: XPE, Definitive Therapy
Arm/Group | Head and Neck Cancer Patients
Started | 37
Completed | 33
Not Completed | 4
Period: Maintenance Cetuximab
Arm/Group | Head and Neck Cancer Patients
Started | 31
Completed | 17
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 55 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants with a best response of complete response or partial response. Disease assessments were based on Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0.
Time Frame: Up to 36 months
Population: Treated with docetaxel 75 mg/m^2 day 1, cisplatin 75 mg/m^2 day 1, and cetuximab 250 mg/m^2 days 1, 8, and 15 (after an initial loading dose of 400 mg/m^2), termed TPE, repeated every 21 days for three cycles.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Head and Neck Cancer Patients: Patients with locally advanced HNC, including squamous and undifferentiated histologies, treated with docetaxel 75 mg/m^2 day 1, cisplatin 75 mg/m^2 day 1, and cetuximab 250 mg/m^2 days 1, 8, and 15 (after an initial loading dose of 400 mg/m^2), termed TPE, repeated every 21 days for three cycles
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 37
percentage of participants | 86 [75 to 98]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: as for outcome 1
Time Frame: Up to 36 months
Population: Docetaxel 75 mg/m^2 day 1, cisplatin 75 mg/m^2 day 1, and cetuximab 250 mg/m^2 days 1, 8, and 15 (after an initial loading dose of 400 mg/m^2), termed TPE, repeated every 21 days for three cycles, followed by radiotherapy with concurrent cisplatin 30 mg/m^2 and cetuximab weekly (XPE).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 33
percentage of participants | 100 [91 to 100]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is an estimated percentage of participants without disease progression at two years (or three years) after the start of study treatment. Progression was defined using Response Evaluation Criteria In Solid Tumors (RECIST), version 1.0. The two-year and three-year PFS ended up being the same in this study.
Time Frame: Up to 36 months
Population: All participants that started were evaluable for this outcome measure, except for the one patient removed from study due to hypersensitivity reaction on cycle 1, day 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 38
percentage of participants
  two-year PFS | 70 [53 to 82]
  three-year PFS | 70 [53 to 82]

4. Secondary Outcome: 2-year Overall Survival (OS)
Description: Two-year OS is an estimated percentage of participants still living at two years after the start of study treatment.
Time Frame: Up to 24 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 38
percentage of participants | 84 [68 to 93]

5. Secondary Outcome: 3-year Overall Survival (OS)
Description: Three-year OS is an estimated percentage of participants still living at three years after the start of study treatment.
Time Frame: Up to 36 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 38
percentage of participants | 74 [54 to 86]

6. Secondary Outcome: Quality of Life (QOL)
Description: Effect of treatment on acute and late QOL and functional status using Functional Assessment of Cancer Therapy-General (FACT-G) with FACT-Head and Neck (FACT-HN) subscale. The instructions to the participant were: "Below is a list of statements that other people with your illness have said are important. By circling one number per line, please indicate how true each statement has been for you during the past 7 days." The choices for each statement ranged from 0 (not at all) to 4 (very much). The FACT-G and FACT-Head and Neck total scores were computed by summing 27 and 39 questions respectively, for four subscales: physical well-being, social well-being, emotional well-being, and functional well-being. Questions for both assessments are phrased so that higher numbers/values indicate a better health state.
Time Frame: Pre-treatment, Post-induction, 3 months after XPE and 12 months after XPE
Population: Analysis was completed using all responses actually obtained.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Head and Neck Cancer Patients
Number analyzed (Participants) | 30
units on a scale
  FACT-G Total Score Pre-treatment | 77.4311 (16.56741)
  FACT-G Total Score Post-induction: number analyzed (Participants) | 22
  FACT-G Total Score Post-induction | 75.6303 (15.68977)
  FACT-G Total Score 3 months after XPE: number analyzed (Participants) | 22
  FACT-G Total Score 3 months after XPE | 71.3864 (17.51042)
  FACT-G Total Score 12 months after XPE: number analyzed (Participants) | 19
  FACT-G Total Score 12 months after XPE | 86.6702 (18.82226)
  FACT-HN Pre-treatment | 25.7000 (6.74230)
  FACT-HN Post-induction: number analyzed (Participants) | 22
  FACT-HN Post-induction | 25.1250 (7.42332)
  FACT-HN 3 months after XPE: number analyzed (Participants) | 22
  FACT-HN 3 months after XPE | 19.4545 (5.01167)
  FACT-HN 12 months after XPE: number analyzed (Participants) | 19
  FACT-HN 12 months after XPE | 24.5263 (7.50088)

7. Other Pre Specified Outcome: EGFR-related Serum Markers
Description: Evaluation of changes in serum markers (EGFR-related) before and after therapy in the above patient population, and expression of pAKT, pMAPK, and other EGFR pathway-related markers as well angiogenesis biomarkers.
Time Frame: Up to 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Head and Neck Cancer Patients
Serious Adverse Events (participants affected / at risk) | 32/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Head and Neck Cancer Patients (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 13
Platelets (Blood and lymphatic system disorders) | 1
Cardiac arrhythmia (Cardiac disorders) | 1
Ocular/Visual - Other (Specify) (Eye disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Hemorrhage, GI, Stomach (Gastrointestinal disorders) | 1
Hemorrhage, GI, Upper GI NOS (Gastrointestinal disorders) | 1
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Rigors/chills (General disorders) | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1
Infection - Other (Specify) (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Glucose, serum-high (hyperglycemia) (Investigations) | 1
Magnesium, serum-low (hypomagnesemia) (Investigations) | 6
Potassium, serum-high (hyperkalemia) (Investigations) | 1
Potassium, serum-low (hypokalemia) (Investigations) | 1
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Pain, Joint (Musculoskeletal and connective tissue disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Pain-Other (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 2
Rash: dermatitis associated with radiation, Radiation (Skin and subcutaneous tissue disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Head and Neck Cancer Patients (N=39)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Febrile neutropenia (unknown origin without documented infection)(ANC <1.0 x 10^9/L) (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 25
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 5
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 1
Lymphatics - Other (Blood and lymphatic system disorders) | 1
Cardiac Arrhythmia - Other (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Atrial flutter (Cardiac disorders) | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 2
Pain, External ear (Ear and labyrinth disorders) | 1
Pain, Middle ear (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Eyelid dysfunction (Eye disorders) | 1
Ocular/Visual - Other (Eye disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 13
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 31
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2
Gastrointestinal - Other (Gastrointestinal disorders) | 6
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemorrhage, GI, Rectum (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 26
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 27
Pain, Abdomen NOS (Gastrointestinal disorders) | 2
Pain, Oral cavity (Gastrointestinal disorders) | 26
Pain, Stomach (Gastrointestinal disorders) | 1
Perforation, GI, Esophagus (Gastrointestinal disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 21
Edema: head and neck (General disorders) | 2
Edema: limb (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 36
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L) (General disorders) | 12
Injection site reaction/extravasation changes (General disorders) | 1
Pain - Other (General disorders) | 10
Pain, Face (General disorders) | 4
Pain, Pain NOS (General disorders) | 3
Rigors/chills (General disorders) | 4
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4
Infection - Other (Infections and infestations) | 3
Infection (documented) with Grade 3 or 4 neutrophils (ANC <1.0 x 10^9/L), Eye NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Joint (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection with unknown ANC, Mucosa (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Creatinine (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 19
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 16
Platelets (Investigations) | 9
Weight loss (Investigations) | 10
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 12
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 23
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Pain, Back (Musculoskeletal and connective tissue disorders) | 1
Pain, Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 1
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain, Joint (Musculoskeletal and connective tissue disorders) | 4
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 3
Pain, Neck (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 5
Neurology - Other (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 16
Pain, Head/headache (Nervous system disorders) | 7
Seizure (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Mood alteration, Agitation (Psychiatric disorders) | 1
Mood alteration, Anxiety (Psychiatric disorders) | 2
Mood alteration, Depression (Psychiatric disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Nose (Respiratory, thoracic and mediastinal disorders) | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis/stomatitis (clinical exam), Esophagus (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis/stomatitis (functional/symptomatic), Esophagus (Respiratory, thoracic and mediastinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic), Trachea (Respiratory, thoracic and mediastinal disorders) | 1
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 5
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 8
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 26
Pain, Skin (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 19
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 8
Rash: dermatitis associated with radiation, Radiation (Skin and subcutaneous tissue disorders) | 13
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No